CLINICAL TRIAL: NCT05787444
Title: Clinical Validation of the LumiraDx SARS-CoV-2 & Flu A/B Test in Anterior Nares Nasal Samples For Point-of-Care (POC) Use
Brief Title: Clinical Validation of the LumiraDx SARS-CoV-2 & Flu A/B Test in Detecting and Differentiating Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2), Influenza A (Flu A), and/or Influenza B (Flu B)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: LumiraDx UK Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: CS-1489-01; 13379 (Other: RADx)
Record Dates: First submitted 2023-03-16; First posted 2023-03-28 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-05

CONDITIONS: SARS-CoV-2; Influenza A; Influenza B; Asymptomatic COVID-19
Keywords: LumiraDx Diagnostic tests; Multiplex SARS-CoV-2; Influenza A; Influenza B; Asymptomatic; COVID-19 Infections; Coronavirus Lung disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Anterior Nasal Swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (1):
- symptomatic: Subject is currently exhibiting fever, or one or more symptoms associated with COVID-19 or influenza (such as, but not limited to, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting or diarrhea) and must present within 6 days of symptom onset. Subject must still be exhibiting symptoms on the day of sample collection.
  Interventions: Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B

INTERVENTIONS:
Diagnostic Test: LumiraDx SARS-CoV-2 & Flu A/B — The LumiraDx SARS-CoV-2 & Flu A/B test is an automated rapid microfluidic immunofluorescence assay for use with the LumiraDx Platform, for near-patient testing, intended for the qualitative and differential detection of nucleocapsid viral antigens from SARS-CoV-2, influenza A, and influenza B in an anterior nares sample (from both nostrils) collected by a healthcare professional for individuals aged 2 years and older. The test is authorized for individuals with symptoms of COVID-19, influenza A and B within the first 6 days of symptom onset.

SUMMARY:
This is a prospective multicenter study conducted to evaluate the performance of the LumiraDx SARS-CoV-2 & Flu A/B tests at point of care sites. Subjects presenting with symptoms suggestive of coronavirus disease 2019 (COVID-19) and Influenza at the time of the study visit will be enrolled and asked to donate swab sample(s) for testing on the device under evaluation.

DETAILED DESCRIPTION:
This will be a prospective study at point of care sites in the United States for the clinical validation of the LumiraDx SARS-CoV-2 & Flu A/B test for the differential detection of the SARS-CoV-2, and influenza A & B using anterior nasal samples. Up to 1,500 or more symptomatic subjects who are currently experiencing symptoms associated with COVID-19 and Influenza A & B may be enrolled.

The samples are obtained from each subject using standard collection methods and are processed and tested by untrained operators without laboratory training and with no prior experience using the candidate test.

The primary objective of this study is to evaluate the performance (positive percent agreement, negative percent agreement and 95% confidence intervals for upper and lower bounds) of the LumiraDx SARS-CoV-2 & Flu A/B test for the qualitative and differential detection of SARS-CoV-2, Influenza A & B virus antigen using anterior nares samples collected by a healthcare professional, compared to a 510(k) cleared or Emergency Use Authorized (EUA) high-sensitivity reverse transcription-polymerase chain reaction (RT-PCR) test for COVID-19 and a 510(k) cleared Influenza A/B test.

The secondary objective is to assess the usability and user accuracy/performance around limit of detection (LoD) of the investigational test using a questionnaire and accuracy study.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to study enrollment.
2. Male or female aged 2 years of age or older
3. Subject is currently exhibiting fever, or one or more symptoms associated with COVID-19 or influenza (such as, but not limited to, chills, cough, shortness of breath or difficulty breathing, fatigue, new loss of taste or smell, sore throat, congestion or runny nose, nausea or vomiting or diarrhea) and must present within 6 days of symptom onset. Subject must still be exhibiting symptoms on the day of sample collection.

Exclusion Criteria:

1. Subject does not understand or is not able and willing to sign the study informed consent or be verbally assented.
2. Subject has had the seasonal influenza and/or the SARS-CoV-2 vaccine within the past 5 days.
3. Subject is not able to tolerate sample collection.
4. Subject is currently undergoing antiviral treatment such as baloxavir marboxil (trade name Xofluza®), oseltamivir (Tamiflu®), zanamivir (Relenza®), and peramivir (Rapivab®).
5. Subjects undergoing treatment currently and/or within the past thirty (30) days with prescription medication to treat novel Coronavirus SARS-CoV-2 infection, which may include but is not limited to Remdesivir (Veklury), Paxlovid, molnupiravir or receiving convalescent plasma therapy for SARS-CoV-2.
6. Subjects who have taken Evusheld (tixagevimab/cilgavimab) within the last 90 days.
7. Subjects who have had a nasal wash or aspirate as part of their standard of care treatment on day of study visit prior to study sample collection.
8. Subjects who have had recent craniofacial injury or surgery, including to correct deviation of the nasal septum, within the previous six (6) months.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The entire population that met the eligibility criteria. Symptomatic subjects who are currently exhibiting fever, or one or more symptoms associated with COVID-19 or influenza and present within 6 days of symptom onset. Subject must still be exhibiting symptoms on the day of sample collection.
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Performance evaluation of the LumiraDx SARS-CoV-2 & Flu A/B in point of care settings | 6 months
  Evaluate the performance of the LumiraDx SARS-CoV-2 & Flu A/B test in detecting and differentiating SARS-CoV-2, influenza A and influenza B in fresh nasal swab specimens from symptomatic patients. Performance will be evaluated by use of statistical analysis techniques to assess negative and positive percent agreement (NPA, PPA) of the LumiraDx test results versus an FDA-approved method where a result of 100% NPA or PPA would equate to complete agreement with the reference method and 0% would equate to no agreement.

SECONDARY OUTCOMES:
Validation of the LumiraDx SARS-CoV-2 & Flu A/B for use by intended users | 2 months
  Each site will conduct testing with contrived samples prepared by the Sponsor in a User Accuracy study. Additionally, each operator will complete a usability questionnaire evaluating various features of the investigational test and instructions. Users will use the Likert scale (strongly agree - strongly disagree) to rate their responses. Results will be collated and assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Randall Quinn, MD, Principal Investigator — Cullman Clinical Trials
Locations (1):
- Cullman Clinical Trials, Cullman, Alabama, United States